CLINICAL TRIAL: NCT03146546
Title: Diagnostic and Prognostic Biomarkers to Elucidate Sepsis Endotypes
Brief Title: STUDY00015328: Sepsis Endotypes
Status: Enrolling by invitation | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Anthony Bonavia, Professor, Penn State Health Milton S Hershey Medical Center
Other Study IDs: 7188
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sepsis: Patients with sepsis as defined by the Sepsis-3 criteria
- Control: Patients without sepsis, as defined by the Sepsis-3 criteria

SUMMARY:
Determine the utility of biomarkers measured in blood and body fluid (stool, saliva, tracheal aspirate) when combined with clinical data, for predicting sepsis phenotypes that are associated with poor clinical outcomes. We hypothesize that resistin is a biomarker which provides critical prognostic information when used in conjunction with standard clinical data, in patients with sepsis and septic shock.

DETAILED DESCRIPTION:
Day 1 Sample Collection: 20ml of blood for chemical and genetic biomarker analysis. ≤1ml of saliva, stool, and tracheal aspirate for inflammatory marker analysis. Quadratus lumborum muscle size measurement and CT abdomen correlation. If not part of routine care, additional blood tests for cell differential, procalcitonin, and inflammatory markers.

Electronic Medical Records (EMR) Data: APACHE II and SOFA severity scores. Demographics, vital signs, inflammatory markers, organ dysfunction markers, and various blood chemistry values.

Days 2-3 Daily Documentation: Record the most abnormal value for the same parameters as Day 1.

Days 3-5 (Once) Sample Collection: Repeat of blood, saliva, stool, and tracheal aspirate collection. EMR data access for severity scores and other clinical parameters.

Days 5-6 Daily Documentation: Continued recording of the most abnormal values for clinical parameters.

Days 7-10 (Once) Sample Collection: Repeat of blood, saliva, stool, and tracheal aspirate collection. Measurement of muscle size and CT correlation. EMR data access for the same parameters as earlier.

Day 14 (or Discharge) Final Sample Collection: 20ml of blood and other samples, with no more than 1 ml/kg of blood collected over the entire study.

EMR and Clinical Data: Collection of severity scores, vital signs, inflammation markers, organ dysfunction markers, and other clinical variables.

Day 30, 3 Months, 6 Months, and 1 Year Long-term Outcomes: EMR review for clinical outcomes such as date of death, re-hospitalization, persistent critical illness. Phone interviews to gather subjective data about the post-hospitalization course and complications.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age ≥ 18 )
2. gender: male or female
3. Cognitively intact or impaired patients, given that sepsis may cause a certain degree of cognitive dysfunction in patients. All patients in the control group (no sepsis) will be cognitively intact
4. Clinical suspicion for sepsis (except for control/comparison group for whom infection is NOT a current concern)

Exclusion Criteria:

1. Patients with hematologic malignancies
2. Pregnant women
3. Patient/surrogate is not fluent in English and no translation services are available
4. Long-term immunosuppressive therapy
5. Prisoner

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients in the intensive care unit (ICU) who meet critera for sepsis, as defined by the Sepsis-3 criteria and who are not excluded by any of the exclusion factors listed in the "Eligibility Criteria".
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
death and chronic critical illness | 5 years for completion of study, 1 year follow up per patient enrolled
  The primary outcome is a composite binary variable consisting of early death and chronic critical illness which we will determine on or before day 14 after sepsis onset.

SECONDARY OUTCOMES:
The expression of BPGM and AP2 transcripts | 5 years for completion of study, 1 year follow up per patient enrolled
  sepsis-associated gene pathways
Clinical variables | 5 years for completion of study, 1 year follow up per patient enrolled
  including demographic variables (eg, age, sex, Elixhauser comorbidities), vital signs (eg, heart rate, respiratory rate, Glasgow Coma Scale score, systolic blood pressure, temperature, and oxygen saturation), markers of inflammation (eg, white blood cell count, premature neutrophil count [also called bands], erythrocyte sedimentation rate, and C-reactive protein), markers of organ dysfunction or injury (eg, alanine aminotransferase, aspartate aminotransferase, total bilirubin, blood urea nitrogen, creatinine, international normalized ratio, partial pressure of oxygen, platelets, and troponin), and serum levels of glucose, sodium, hemoglobin, chloride, bicarbonate, lactate, and albumin.
Acute Physiology and Chronic Health Evaluation II Score | 5 years for completion of study, 1 year follow up per patient enrolled
  scale 0-71, with higher scores being worse
Sequential Organ Failure Assessment | 5 years for completion of study, 1 year follow up per patient enrolled
  scale of 0-24, with higher scores being worse score
Muscle measurements | 5 years for completion of study, 1 year follow up per patient enrolled
  Clinical measurement of quadriceps depth (ultrasound) and skeletal muscle area (on existing CT scan)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bonavia, M.D., Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kovach MA, Standiford TJ. The function of neutrophils in sepsis. Curr Opin Infect Dis. 2012 Jun;25(3):321-7. doi: 10.1097/QCO.0b013e3283528c9b. PMID 22421753
- [Background] Stephan F, Yang K, Tankovic J, Soussy CJ, Dhonneur G, Duvaldestin P, Brochard L, Brun-Buisson C, Harf A, Delclaux C. Impairment of polymorphonuclear neutrophil functions precedes nosocomial infections in critically ill patients. Crit Care Med. 2002 Feb;30(2):315-22. doi: 10.1097/00003246-200202000-00009. PMID 11889301
- [Background] Delano MJ, Thayer T, Gabrilovich S, Kelly-Scumpia KM, Winfield RD, Scumpia PO, Cuenca AG, Warner E, Wallet SM, Wallet MA, O'Malley KA, Ramphal R, Clare-Salzer M, Efron PA, Mathews CE, Moldawer LL. Sepsis induces early alterations in innate immunity that impact mortality to secondary infection. J Immunol. 2011 Jan 1;186(1):195-202. doi: 10.4049/jimmunol.1002104. Epub 2010 Nov 24. PMID 21106855
- [Background] Cummings CJ, Martin TR, Frevert CW, Quan JM, Wong VA, Mongovin SM, Hagen TR, Steinberg KP, Goodman RB. Expression and function of the chemokine receptors CXCR1 and CXCR2 in sepsis. J Immunol. 1999 Feb 15;162(4):2341-6. PMID 9973513
- [Background] Macdonald SP, Stone SF, Neil CL, van Eeden PE, Fatovich DM, Arendts G, Brown SG. Sustained elevation of resistin, NGAL and IL-8 are associated with severe sepsis/septic shock in the emergency department. PLoS One. 2014 Oct 24;9(10):e110678. doi: 10.1371/journal.pone.0110678. eCollection 2014. PMID 25343379
- [Background] Koch A, Gressner OA, Sanson E, Tacke F, Trautwein C. Serum resistin levels in critically ill patients are associated with inflammation, organ dysfunction and metabolism and may predict survival of non-septic patients. Crit Care. 2009;13(3):R95. doi: 10.1186/cc7925. Epub 2009 Jun 19. PMID 19545363
- [Background] Sunden-Cullberg J, Nystrom T, Lee ML, Mullins GE, Tokics L, Andersson J, Norrby-Teglund A, Treutiger CJ. Pronounced elevation of resistin correlates with severity of disease in severe sepsis and septic shock. Crit Care Med. 2007 Jun;35(6):1536-42. doi: 10.1097/01.CCM.0000266536.14736.03. PMID 17452927
- [Background] Singbartl K, Miller L, Ruiz-Velasco V, Kellum JA. Reversal of Acute Kidney Injury-Induced Neutrophil Dysfunction: A Critical Role for Resistin. Crit Care Med. 2016 Jul;44(7):e492-501. doi: 10.1097/CCM.0000000000001472. PMID 26646460